CLINICAL TRIAL: NCT00012311
Title: Multi-Cycle High-Dose Chemotherapy Versus Optimized Conventionally-Dosed Chemotherapy in Patients With Metastatic Breast Cancer: A Phase II Prospective Randomized Trial
Brief Title: Chemotherapy Plus Peripheral Stem Cell Transplantation Compared With Chemotherapy Alone in Treating Women With Stage IV Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068504; CPMC-IRB-9244; NCI-G01-1922
Record Dates: First submitted 2001-03-03; First posted 2004-04-13 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2001-09

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; CMF regimen; Carboplatin; Cyclophosphamide; Docetaxel; Doxorubicin; Etoposide; Fluorouracil; Ifosfamide; Methotrexate; Thiotepa; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: CMF regimen
Drug: carboplatin
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: fluorouracil
Drug: ifosfamide
Drug: methotrexate
Drug: thiotepa
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. It is not yet known if chemotherapy followed by peripheral stem cell transplantation is more effective than chemotherapy alone in treating metastatic breast cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of combination chemotherapy plus peripheral stem cell transplantation with that of chemotherapy alone in treating women who have stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of multi-course high-dose chemotherapy with autologous peripheral blood stem cell transplantation versus standard-dose chemotherapy in women with metastatic breast cancer. II. Compare the five year event-free survival, in terms of time to progression or time to death due to toxic effects, in patients treated with these regimens. III. Compare the response rate and overall survival of patients treated with these regimens. IV. Compare the toxicity of these regimens in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms. Arm I: Patients receive docetaxel and doxorubicin once followed by filgrastim (G-CSF) daily for approximately 1 week. Treatment repeats approximately every 3 weeks for 4 courses. Patients then receive cyclophosphamide, methotrexate, and fluorouracil on days 7 and 8 every 4 weeks for 4 courses. Arm II: Patients receive docetaxel, doxorubicin, and G-CSF as in arm I for 3 courses. Patients undergo leukapheresis daily for 3 or 4 days. Patients then receive 1 course of ifosfamide, etoposide, and carboplatin daily for 4 days when blood counts recover, followed by 1 course of cyclophosphamide and thiotepa daily for 4 days. Patients undergo peripheral blood stem cell reinfusion following each course.

PROJECTED ACCRUAL: A total of 264 patients (132 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage IV breast carcinoma Bone metastasis as only form of metastatic disease allowed No evidence of bone marrow involvement by aspirate or biopsy No brain metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 to 59 Sex: Female Menopausal status: Not specified Performance status: Karnofsky 80-100% Life expectancy: More than 3 months Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 9 g/dL PT normal Activated PTT normal Hepatic: Bilirubin normal (unless benign congenital hyperbilirubinemia is present) No AST/ALT greater than 1.5 times upper limit of normal (ULN) together with alkaline phosphatase greater than 2.5 times ULN No active hepatitis B or C Renal: Creatinine normal Cardiovascular: Ejection fraction normal by MUGA or echocardiogram No active heart disease No prior myocardial infarction or other manifestation of coronary artery disease Other: More than 1,000 calories/day oral intake HIV negative No active serious medical or psychiatric disease No other prior or concurrent malignancy except basal cell skin cancer or carcinoma in situ of the cervix No allergy to polysorbate 80 or E. coli-derived products No peripheral neuropathy greater than grade 2 Not pregnant Negative pregnancy test

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for metastatic disease No prior mitomycin, nitrosoureas, or platinum coordination complexes Prior adjuvant chemotherapy allowed if completed more than 6 months prior to relapse with metastases No more than 300 mg/m2 prior doxorubicin or 450 mg/m2 prior epirubicin Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to the brain or marrow-bearing pelvis Prior radiotherapy to lower pelvis allowed if the upper border of the radiotherapy field is below the upper border of the acetabulum No other prior radiotherapy to the pelvis Surgery: At least 2 weeks since prior major surgery Other: No other concurrent anti-cancer therapy

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: Linda T. Vahdat, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center, New York, New York, United States